CLINICAL TRIAL: NCT02494141
Title: Curcumin Therapy to Treat Vascular Dysfunction in Children and Young Adults With ADPKD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15-0902
Record Dates: First submitted 2015-06-25; First posted 2015-07-10 (Estimated); Results first posted 2022-03-03 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: Polycystic Kidney, Autosomal Dominant
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant | interventions — Curcumin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Curcumin (Experimental): 25/mg/kg per day for 1 year.
  Interventions: Drug: Curcumin
- Placebo (Placebo Comparator): Equivalent placebo for 1 year.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Curcumin — Dietary Supplement
  Other Names: Longvida
  Arms: Curcumin
Other: Placebo
  Arms: Placebo

SUMMARY:
The proposed research will determine the effectiveness of curcumin for improving the health and function of arteries in children and young adults with autosomal dominant polycystic kidney disease (ADPKD). The study also will provide insight into how curcumin improves artery health by determining the physiological mechanisms (biological reasons) involved and offer exploratory evidence if curcumin can slow kidney growth. This will be done by comparing these measurements in children and young adults who are randomized to receive either curcumin or placebo for 1 year.

DETAILED DESCRIPTION:
Although often considered to be a disease of adults, complications of autosomal dominant polycystic kidney disease (ADPKD) begin in childhood. While ADPKD causes the continued growth of multiple kidney cysts that ultimately result in loss of kidney function, the leading cause of death among patients with ADPKD is cardiovascular disease. Treatment options to prevent cardiovascular disease in adults with ADPKD are limited, thus childhood may be an important time to reduce risk. Curcumin is a safe, naturally occurring substance found in the Indian spice tumeric, which is in curry powder. The proposed research will determine the effectiveness of curcumin for improving the health and function of arteries in children and young adults with ADPKD. The study also will provide insight into how curcumin improves artery health by determining the physiological mechanisms (biological reasons) involved and offer exploratory evidence if curcumin can slow kidney growth. This will be done by comparing these measurements in children and young adults who are randomized to receive either curcumin or placebo for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* ADPKD diagnosis
* Normal renal function (estimated glomerular filtration rate >80 mL/min/1.73m^2)
* Ability to provide informed consent

Exclusion Criteria:

* Currently taking a curcumin supplement
* Current smoking or history of smoking in the past 12 months
* Marijuana use within 2 weeks prior to FMDBA and aPWV testing
* Antioxidantand/or omega-3 fatty acid use within the past 4 weeks prior to FMDBA and aPWV testing and for the duration of the study
* Alcohol dependence and abuse
* History of hospitalization within the last 3 months
* Active infection or antibiotic therapy
* Pregnancy, lactation, or unwillingness to use adequate birth control
* Body-mass index >95th percentile in ages 6-17 or >40 kg/m2 in ages 18-25
* Inability to cooperate with/clinical contraindication for MRI including severe claustrophobia, implants, devices, or non-removable body piercings

Ages: 6 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 68 (Actual)
Dates: Start 2015-11-12 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristen L Nowak, Ph.D., Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in ADPKD. Data shared will be coded, with no PHI included. Approval of the request and execution of all applicable agreements (i.e. data use agreement) are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, ICF
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA).

REFERENCES:
- [Derived] Nowak KL, Farmer-Bailey H, Wang W, You Z, Steele C, Cadnapaphornchai MA, Klawitter J, Patel N, George D, Jovanovich A, Soranno DE, Gitomer B, Chonchol M. Curcumin Therapy to Treat Vascular Dysfunction in Children and Young Adults with ADPKD: A Randomized Controlled Trial. Clin J Am Soc Nephrol. 2022 Feb;17(2):240-250. doi: 10.2215/CJN.08950621. Epub 2021 Dec 14. PMID 34907021

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Equivalent placebo for 1 year.
  Placebo
Period: Overall Study
Arm/Group | Curcumin | Placebo
Started | 34 | 34
Completed | 28 | 29
Not Completed | 6 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Curcumin | Placebo | Total
Number analyzed (Participants) | 34 | 34 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 18 (6) | 19 (5) | 18 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 18 | 37
  Male | 15 | 16 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 6
  Not Hispanic or Latino | 32 | 30 | 62
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 33 | 32 | 65
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 34 | 34 | 68
Estimated Glomerular Filtration Rate [Mean (Standard Deviation); unit: ml/minute/1.73m^2] — Measure of kidney function. A score of about 100 would mean that kidneys are functioning properly. Lower scores mean lower function, and a worse outcome.
  ml/minute/1.73m^2 | 115 (16) | 118 (19) | 117 (17)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Brachial Artery Flow-mediated Dilation (FMD-BA)
Description: co-primary endpoint
Time Frame: Baseline, Month 12
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | Curcumin | Placebo
Number analyzed (Participants) | 34 | 34
percent change | 1.14 [-0.84 to 3.13] | 0.3 [-1.34 to 2.00]

2. Primary Outcome: Change in Aortic Pulse-wave Velocity (aPWV) (cm/Sec)
Description: co-primary endpoint
Time Frame: Baseline, Month 12
Measure: Mean (95% Confidence Interval); unit: cm/sec
Arm/Group | Curcumin | Placebo
Number analyzed (Participants) | 34 | 34
cm/sec | 0.6 [-25.7 to 26.9] | 6.5 [-20.4 to 33.5]

3. Secondary Outcome: Change in Urinary 8-iso-prostaglandin F2α (8-isoprostane)
Description: Urine marker of oxidative stress. Values are normalized to urinary creatinine.
Time Frame: Baseline, Month 12
Population: Some participants were excluded because 12 month data was not collected.
Measure: Mean (95% Confidence Interval); unit: mg/dl
Arm/Group | Curcumin | Placebo
Number analyzed (Participants) | 28 | 29
mg/dl | 0.00 [-0.34 to 0.34] | 0.27 [-0.14 to 0.69]

4. Secondary Outcome: Change in C-reactive Protein
Description: Circulating marker of inflammation
Time Frame: Baseline, Month 12
Population: Some participants were excluded because their 12 month data was not collected.
Measure: Mean (95% Confidence Interval); unit: mg/L
Arm/Group | Curcumin | Placebo
Number analyzed (Participants) | 27 | 29
mg/L | 0.21 [-0.47 to 0.88] | 0.17 [-0.36 to 0.70]

5. Secondary Outcome: Change in Interleukin-6
Description: Circulating marker of inflammation
Time Frame: Baseline, Month 12
Population: Some participants were excluded because 12 month data was not collected.
Measure: Mean (95% Confidence Interval); unit: picograms/mL
Arm/Group | Curcumin | Placebo
Number analyzed (Participants) | 27 | 29
picograms/mL | 2.24 [1.69 to 2.80] | 2.33 [1.89 to 2.76]

6. Secondary Outcome: Percent Change in Oxidative Stress-associated Suppression of Endothelium-dependent Dilation (EDD)
Description: The influence of oxidative stress on FMD-BA will be determined by infusing a supraphysiological dose of ascorbic acid known to scavenge superoxide or isovolumic saline. The outcome measure describes the value of the percent change with ascorbic acid compared to saline observed at baseline and the value of the percent change with ascorbic acid compared to saline at the month 12 timepoint.
Time Frame: Baseline, Month 12
Population: This outcome measure was only collected for a subgroup of participants
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Curcumin | Placebo
Number analyzed (Participants) | 12 | 12
Percent change
  Baseline | 3.0 (0.95) | 1.7 (3.0)
  Month 12 | 1.1 (3.5) | 1.4 (2.6)

7. Secondary Outcome: Change in Oxidative Stress-Associated Suppression of Large Elastic Artery Stiffness
Description: The influence of oxidative stress on aPWV will be determined by infusing a supraphysiological dose of ascorbic acid known to scavenge superoxide or isovolumic saline.
Time Frame: Baseline, Month 12
Population: This outcome measure was not collected for any participants.
Arm/Group | Curcumin | Placebo
Number analyzed (Participants) | 0 | 0

8. Other Pre Specified Outcome: Change in Alanine Transaminase (ALT )
Description: Liver enzymes will be monitored for safety.
Time Frame: month 1, 6, and 12
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Change in Aspartate Aminotransferase (AST)
Description: Liver enzymes will be monitored for safety.
Time Frame: month 1, 6, and 12
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Change in Height-corrected Total Kidney Volume
Description: Total kidney volume will be measured by MRI
Time Frame: Baseline, Month 12
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 12 Months
Description: Rows listed to include multiple adverse events (i.e., "Flatulence, constipation, diarrhea, or nausea") were monitored/assessed in this manner.
Arm/Group | Curcumin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/34
Other Adverse Events (participants affected / at risk) | 15/34 | 9/34
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Curcumin (N=34) | Placebo (N=34)
Gastrointestinal issues (Gastrointestinal disorders) | 7 (7) | 7 (7) — Flatulence, constipation, diarrhea, or nausea
Warming or redness of face (Vascular disorders) | 2 (2) | 0 (0)
Tingling of tongue/mouth (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Headache (General disorders) | 1 (1) | 1 (1)
Dry Mouth (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Eye redness, dryness, or swelling (Eye disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-03-12): https://cdn.clinicaltrials.gov/large-docs/41/NCT02494141/Prot_SAP_000.pdf
  • Informed Consent Form (2020-12-11): https://cdn.clinicaltrials.gov/large-docs/41/NCT02494141/ICF_001.pdf